CLINICAL TRIAL: NCT04002141
Title: Assessment and Prevention of Pain During Ovarian Stimulation in Patients With Endometriosis
Acronym: APPOSE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18-26544
Record Dates: First submitted 2019-05-28; First posted 2019-06-28 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Endometriosis; Ovarian Hyperstimulation
Keywords: Endometriosis; Letrozole
MeSH Terms: conditions — Endometriosis | interventions — Letrozole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Endometriosis Letrozole (Experimental): Participants will be asked to take 5mg letrozole daily throughout their ovarian stimulation and for 2 weeks following retrieval. Participants will be blinded to their randomization to letrozole. Participants will be asked to complete surveys during their stimulation and up to 12 weeks following retrieval to evaluate endometriosis associated symptoms. Specifically, surveys will be administered at baseline ultrasound appointment for controlled ovarian hyperstimulation cycle, the day of trigger shot, 3 weeks following egg retrieval, 6 weeks following egg retrieval and 12 weeks following egg retrieval. There will be a total of 20 participants in this arm.
  Interventions: Drug: Letrozole
- Endometriosis Placebo (Placebo Comparator): Participants will be asked to take one tablet placebo daily throughout their ovarian stimulation and for 2 weeks following retrieval. Participants will be blinded to their randomization to placebo. Participants will be asked to complete surveys during their stimulation and up to 12 weeks following retrieval to evaluate endometriosis associated symptoms. Specifically, surveys will be administered at baseline ultrasound appointment for controlled ovarian hyperstimulation cycle, the day of trigger shot, 3 weeks following egg retrieval, 6 weeks following egg retrieval and 12 weeks following egg retrieval. There will be a total of 20 participants in this arm.
  Interventions: Drug: Placebo oral tablet
- No Endometriosis Control (No Intervention): Participants will be asked to complete surveys during their ovarian stimulation and up to 12 weeks following retrieval to evaluate symptoms of pelvic pain. Specifically, surveys will be administered at baseline ultrasound appointment for controlled ovarian hyperstimulation cycle, the day of trigger shot, 3 weeks following egg retrieval, 6 weeks following egg retrieval and 12 weeks following egg retrieval. There will be a total of 20 participants in this arm.

INTERVENTIONS:
Drug: Placebo oral tablet — 1 tablet oral daily
  Arms: Endometriosis Placebo
Drug: Letrozole — 5mg oral daily
  Arms: Endometriosis Letrozole

SUMMARY:
Randomized double blinded placebo-controlled trial to evaluate the impact of ovarian hyperstimulation on endometriosis-related symptoms and to evaluate the impact of letrozole use during ovarian hyperstimulation with respect to endometriosis-related symptoms, embryo/egg quality and quantity, and pregnancy rates.

DETAILED DESCRIPTION:
Randomized double blinded placebo-controlled trial to evaluate: (1) the impact of letrozole use during ovarian hyperstimulation with respect to endometriosis-related symptoms, embryo/egg quality and quantity, and pregnancy rates, (2) the impact of ovarian hyperstimulation on endometriosis-related symptoms.

There will be a total of 60 participants, 20 participants with endometriosis randomized to the placebo group, 20 participants with endometriosis randomized to the letrozole group and 20 control patients with no history of endometriosis. Letrozole and placebo medication will be started on the first day of gonadotropin injections and continued until the day of trigger shot. Medication will be restarted the night of egg retrieval and continued for 2 weeks post retrieval. Endometriosis associated symptoms will be evaluated using a survey modeled after the clinical survey developed by the World Endometriosis Research Foundation Endometriosis Phenome and Biobanking Harmonisation Project. Surveys will be administered at baseline ultrasound appointment for controlled ovarian hyperstimulation cycle, the day of trigger shot, 3 weeks following egg retrieval, 6 weeks following egg retrieval and 12 weeks following egg retrieval.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-42 years
* Planning to undergo controlled ovarian hyperstimulation
* Prior diagnosis of endometriosis by one of the following: (1) surgical diagnosis (2) endometrioma on pelvic ultrasound
* Planning to freeze all retrieved oocytes/embryos prior to transfer

Exclusion Criteria:

* Hypersensitivity to letrozole
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow-up, or interpretation of study results

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2025-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelle I Cedars, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Center for Reproductive Health, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Endometriosis Letrozole | Endometriosis Placebo | No Endometriosis Control
Started | 20 | 20 | 20
Completed | 20 | 20 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Endometriosis Letrozole | Endometriosis Placebo | No Endometriosis Control | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 20 | 60
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 20 | 60
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Average Delta in Endometriosis Pain Score Pre and Post Stimulation With and Without Use Of Letrozole
Description: To evaluate how letrozole impacts pain scores throughout controlled ovarian hyperstimulation in patients with endometriosis. Pain scores will be evaluated using a 0-10 visual acuity scale, where 0 is no pain and 10 is the worst imaginable pain. The average delta between pre-stimulation pain score and day of trigger shot pain score will be compared between patients with endometriosis receiving placebo and with endometriosis receiving letrozole.
Time Frame: Baseline ultrasound (day 2 of menstrual cycle) and day 12 (average day of trigger shot).
Population: only includes those who completed stimulation and filled out survey for baseline and trigger pain
Measure: Mean (Standard Deviation); unit: Change in score on a scale
Arm/Group | Endometriosis Letrozole | Endometriosis Placebo
Number analyzed (Participants) | 17 | 16
Change in score on a scale | -2.5 (3.9) | -2.7 (3.9)

2. Secondary Outcome: Average Delta in Endometriosis Pain Score Pre and Post Stimulation of Patients Receiving Placebo Compared to No Endometriosis
Description: To evaluate the impact of endometriosis on pain scores throughout controlled ovarian hyperstimulation. Pain scores will be evaluated using a 0-10 visual acuity scale, where 0 is no pain and 10 is the worst imaginable pain. The average delta between pre-stimulation pain score and day of trigger shot will be compared between patients with endometriosis receiving placebo and patients without endometriosis.
Time Frame: Baseline ultrasound (day 2 of menstrual cycle) and day 12 (average day of trigger shot).
Population: only includes those who completed stimulation and filled out surveys for baseline and trigger
Measure: Mean (Standard Deviation); unit: Change in score on a scale
Arm/Group | Endometriosis Placebo | No Endometriosis Control
Number analyzed (Participants) | 16 | 16
Change in score on a scale | -2.7 (3.9) | -0.6 (4.1)

3. Secondary Outcome: Comparative Trends in Endometriosis Pain Score Pre and Post Stimulation of Patients With Endometriosis Receiving Either Placebo or Letrozole and Patients Without Endometriosis
Description: To evaluate the impact of letrozole on endometriosis pain scores throughout controlled ovarian hyperstimulation. Pain scores will be evaluated using a 0-10 visual acuity scale, where 0 is no pain and 10 is the worst imaginable pain. The calculated change in pain scores from pre-stimulation through 12 weeks post retrieval will be compared between patients with endometriosis receiving placebo, patients with endometriosis receiving letrozole and patients without endometriosis.
Time Frame: Pre-stimulation through 12 weeks post retrieval. This time span varies per each patient's course of treatment but is typically 14 weeks in tota
Population: only includes those who filled out baseline and 12 week surveys and completed stimulation
Measure: Mean (Standard Deviation); unit: Change in score on a scale
Arm/Group | Endometriosis Letrozole | Endometriosis Placebo | No Endometriosis Control
Number analyzed (Participants) | 12 | 15 | 15
Change in score on a scale | -0.7 (2.0) | -1.0 (2.3) | -0.6 (2.9)

4. Secondary Outcome: Does Letrozole Impact Egg Quantity in Endometriosis Patients
Description: To describe the impact of letrozole on egg quantity in patients with endometriosis receiving letrozole and those with endometriosis not receiving letrozole and those without endometriosis during controlled ovarian stimulation. The total arm aggregate number of MII eggs retrieved per baseline arm aggregate Antral Follicle Count will be compared between the three groups.
Time Frame: Baseline ultrasound (day 2 of menstrual cycle) and day 14 (average day of egg retrieval).
Population: Only includes those who either froze eggs or used ICSI for fertilization as MII rates are not available for those who used conventional insemination
Measure: Mean (Standard Deviation); unit: percentage of MII grade eggs per AFC
Arm/Group | Endometriosis Letrozole | Endometriosis Placebo | No Endometriosis Control
Number analyzed (Participants) | 16 | 16 | 18
percentage of MII grade eggs per AFC | 0.84 (0.43) | 0.88 (0.44) | 0.73 (0.27)

5. Secondary Outcome: Follicular Fluid
Description: To compare follicular fluid average estradiol levels between placebo, letrozole and control groups.
Time Frame: Baseline ultrasound (day 2 of menstrual cycle) and day 14 (average day of egg retrieval).
Reporting Status: Not Posted

6. Secondary Outcome: Pregnancy Outcomes
Description: To compare pregnancy rates in the placebo, letrozole and control groups. Pregnancy will be defined as positive serum hCG after transfer of embryo. The rate will determined by positive hCG per transfer.
Time Frame: Up to 2 years.
Reporting Status: Not Posted

7. Secondary Outcome: Egg Maturity
Description: To describe the impact of letrozole on egg maturity. Measured by number of MII eggs per total number eggs retrieved in patients with endometriosis receiving letrozole and those with endometriosis not receiving letrozole during controlled ovarian stimulation.
Time Frame: Baseline ultrasound to time of cryopreservation of eggs/embryos, which occurs within 7 days of retrieval..
Reporting Status: Not Posted

8. Secondary Outcome: Embryo Grade
Description: To describe the impact of letrozole on embryo quality. Measured by the average total number of freezable quality embryos (6c or greater, grades 1-2 for symmetry and fragmentation) in patients with endometriosis receiving letrozole and those with endometriosis not receiving letrozole and those without endometriosis during controlled ovarian stimulation.
Time Frame: 2 weeks
Population: only those who completed cycles and froze embryos (does not include egg freezers)
Measure: Mean (Standard Deviation); unit: count of freezable embryos
Arm/Group | Endometriosis Letrozole | Endometriosis Placebo | No Endometriosis Control
Number analyzed (Participants) | 13 | 15 | 9
count of freezable embryos | 2.9 (2.4) | 2.9 (2.4) | 3.3 (2.5)

ADVERSE EVENTS:
Time Frame: Ovarian stimulation baseline through 12 weeks post retrieval. This time span varies per each patient's course of treatment but is typically 14 weeks in tota
Arm/Group | Endometriosis Letrozole | Endometriosis Placebo | No Endometriosis Control
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endometriosis Letrozole (N=20) | Endometriosis Placebo (N=20) | No Endometriosis Control (N=20)
Heavy Vaginal Bleeding (Reproductive system and breast disorders) | 1 (1) | NA | NA — Unanticipated. Possibly Related. Resolved. Heavy vaginal bleeding is not a known side effect of the study medication (letrozole). This event was likely related to pre-existing conditions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT04002141/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-21): https://cdn.clinicaltrials.gov/large-docs/41/NCT04002141/ICF_002.pdf